CLINICAL TRIAL: NCT01443221
Title: Open-label, Randomized, Single-dose, 2-way Crossover Study to Investigate Safety and Pharmacokinetics of Mitiglinide and Metformin in Free Combination and Fixed-dose Combination in Healthy Male Subjects.
Brief Title: Pharmacokinetics of Mitiglinide and Metformin in Free Combination and Fixed-dose Combination in Healthy Male Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CWP-KAD-05
Record Dates: First submitted 2011-09-27; First posted 2011-09-29 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2010-10

CONDITIONS: Healthy
Keywords: mitiglinide; metformin; Pharmacokinetics; Safety
MeSH Terms: interventions — mitiglinide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Free combination (Active Comparator): Free combination of Mitiglinide 10mg and Metformin 500mg
  Interventions: Drug: mitiglinide and metformin
- Fixed-dose combination (Experimental): Fixed-dose combination of Mitiglinide 10mg and Metformin 500mg
  Interventions: Drug: mitiglinide and metformin

INTERVENTIONS:
Drug: mitiglinide and metformin — Free combination of Mitiglinide 10mg and Metformin 500mg
  Arms: Free combination
Drug: mitiglinide and metformin — Fixed-dose combination of Mitiglinide 10mg and Metformin 500mg
  Arms: Fixed-dose combination

SUMMARY:
To investigate safety and pharmacokinetics of mitiglinide and metformin in a fixed-dose combination of mitiglinide/metformin, compared with free combination of mitiglinide and metformin in healthy male subjects.

DETAILED DESCRIPTION:
The Korean clinical practice guidelines on DM recommend that a second oral agent with a different mechanism of action be combined to the regimen when adequate glycemic control is difficult to achieve with an oral hypoglycemic agent accompanied dietary therapy. Therefore, a concurrent administration of metformin, a inhibitor of gluconeogenesis, and mitiglinide, an insulin secretagogue, could be an effective and ideal regimen for management of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Subject with adequate clinical laboratory test results (hematology, blood chemistry, serology, drug abuse, urinalysis etc.)
* Subject with normal results in blood pressure, pulse, body temperature and ECG test
* Subject with body mass index (BMI) between 18.5 kg/m2 and to 25 kg/m2

Exclusion Criteria:

* Clinically significant functional disorder or acute disease
* Chronic disease affecting the absorption, metabolism or excretion of drug
* Any study drug administration within 90 days before the first drug administration
* Use of medicine affecting drug metabolism (inhibition, induction) such as barbital, within 30 days before the first drug administration

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Compare the pharmacokinetic profiles(Cmax, AUClast) of fixed-dose combination versus free dose combination in healthy volunteers | Up to 36 hours postdose for each period

SECONDARY OUTCOMES:
Compare the pharmacokinetic profiles(tmax, t1/2, AUC0-∞) of fixed-dose combination versus free dose combination in healthy volunteers | Up to 36hours postdose for each period

CONTACTS AND LOCATIONS:
Overall Officials: Wooseong Hur, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea